CLINICAL TRIAL: NCT03695289
Title: Adaptation of an Evidence-based Interactive Obesity Treatment Approach (iOTA) for Obesity Prevention in Serious Mental Illness
Brief Title: Interactive Obesity Treatment Approach (iOTA) for Obesity Prevention in Serious Mental Illness
Acronym: iOTA-SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201806118
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Mentally Ill Persons
Keywords: Antipsychotics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iOTA-SMI (Experimental): Participants randomized to iOTA-SMI arm will participate in a 16 week interactive obesity treatment approach (iOTA) program approach.
  Interventions: Behavioral: iOTA SMI
- Health Education Control (Active Comparator): Participants randomized to the Health Education Control arm will receive monthly in-person health coaching visits for 16 weeks.
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: iOTA SMI — Participants randomized to the iOTA SMI arm will undergo an assessment of individual behavior risks, will participate in collaborative goal-setting with a health coach, and will use an interactive text system that will provide ongoing support and self-monitoring of behavior change goals.
  Arms: iOTA-SMI
Behavioral: Health Education Control — Participants randomized to the Health Education Control arm will receive monthly counseling on energy balance, physical activity and nutrition.
  Arms: Health Education Control

SUMMARY:
The proposed project aims to pilot and adapt a scalable and sustainable interactive obesity treatment approach (iOTA) program for adults with serious mental illness (SMI). The project consists of 2 arms: the iOTA SMI arm and the Health Education Control Group arm. The investigators hypothesize that participants in the iOTA intervention group will show favorable change in BMI compared to participants in the Health Education Control group, and participants in the iOTA intervention group will show favorable change in self efficacy with respect to healthy eating and activity compared to those in the Health Education Control group.

DETAILED DESCRIPTION:
Obesity is highly prevalent among chronically-treated individuals with severe mental illness (SMI), exceeding general population rates and contributing to type 2 diabetes, cardiovascular disease (CVD) and premature mortality. Behavioral interventions to reverse obesity in chronic SMI have shown limited effectiveness. There are currently no FDA-approved pharmacotherapies for obesity in SMI, and off-label pharmacotherapies used for weight loss are associated with limited effectiveness or serious adverse event risks. Prior obesity interventions for SMI have often been designed for delivery by existing community mental health center (CMHC) caseworkers/staff. However, mental health workers commonly perceive themselves as overworked and/or career-specialized for psychological rather than medical care, creating barriers to sustainable provider engagement.

Using a design-for-dissemination approach, initial development of the intervention under study incorporated trained health coaches using scalable, inexpensive technology to increase intervention engagement, effectiveness, sustainable reach and cost-effectiveness. Derived from the effective lifestyle intervention used in the Diabetes Prevention Program, the initial parent Interactive Obesity Treatment Approach (iOTA) intervention targets diet, activity and medication adherence, incorporating electronic (e.g., web-based) and interpersonal health coach support. That parent iOTA produces weight loss at 24 months in low-income, racially diverse, community health center populations with obesity, and became a platform for further adaptations of iOTA interventions for other populations and environments, targeting low-income populations with limited web and computer access. Using a formal evaluation process and implementation science framework, the parent iOTA intervention was subsequently adapted to low-income workplace environments, (the Working for You or WfY study, RO1 DK103760; PI: Evanoff) amplifying face-to-face health coach and peer interactions with interactive, semi-automated SMS text messaging, a highly utilized technology among low-income populations.

The investigators further adapted the WfY iOTA for use in adults with chronic SMI using Innovation Corps (I-Corps) methods. Created by the National Science Foundation (NSF) and supported by NIH (PA-18-314), I-Corps uses the Lean Launchpad approach developed by serial entrepreneurs at Stanford for translating academic innovation into practice. The emphasis is on immediate and iterative elicitation of stakeholder feedback via focus groups or short interviews. Using stakeholder input, investigators revise assumptions and hypotheses, testing redesigned offerings and making adjustments to ideas that are not working. In conducting our interviews, we identified "customer" specific (e.g. client, clinician and administrator) barriers to implementation of an un-adapted iOTA in mental health treatment centers. Themes that consistently emerged were concern about limited human resources and added work burden not directly related to the mental health of clients, while clients expressed a desire for more in-person and telephonic coaching time, in addition to text messaging.

Now, the investigators propose to use an overarching treatment adaptation framework18 to further refine our treatment to be more readily implementable for individuals with chronic SMI treated in the CMHC setting. Reproducible adaptation of effective interventions to new target populations and settings requires a formal evaluation process and an implementation science framework. Our overarching aim for this application is to pilot and iteratively adapt a scalable and sustainable iOTA for adults with SMI, planning for future effectiveness testing in a well-powered randomized controlled trial (RCT), and eventual large scale dissemination and implementation.

Aim 1: Conduct a randomized pilot and feasibility study of iOTA-SMI in a diverse sample of adults with chronic SMI, comparing iOTA-SMI to a health education control condition. iOTA-SMI will be piloted in a representative sample of 40 adults ages 18-60 with SMI, randomizing participants 2:1 to 16 weeks of iOTA-SMI versus monthly health education. We hypothesize favorable differences in BMI for iOTA-SMI compared to control. Secondary analyses will assess iOTA effects on health self-efficacy, exploring the relationship between effects on Body Mass Index (BMI) and the target mechanism.

Aim 2: Evaluate feasibility and acceptability of iOTA implementation, making iterative adaptations based on data collected during the pilot. Feasibility, engagement and implementation challenges will be characterized, measured by i) enrollment and retention, ii) obesity intervention acceptability, iii) text response rates, iv) visit adherence v) client expectations, vi) fidelity and vii) CMHC staff-rated acceptability, appropriateness and burden.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60 years
* BMI ≥ 28
* have a diagnosis of a severe and persistent mental illness
* psychiatric symptoms present for at least 6 months prior to screening
* at least 6 months of lifetime antipsychotic exposure prior to screening
* not taking weight loss medications or participating in another behavioral weight loss intervention
* enrolled in case management services
* able to provide written informed consent

Exclusion Criteria:

* acute suicidality at time of screening
* active substance use disorder diagnosis
* unable or unwilling to provide written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 16 Weeks
  Weight in kilograms and height in meters will be measured and combined to calculate BMI in kg/mˆ2 at baseline and following 16 weeks of participation in either an Interactive Obesity Treatment Approach (iOTA) program or a Health Education Program.

CONTACTS AND LOCATIONS:
Overall Officials: Ginger E Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Correll CU, Druss BG, Lombardo I, O'Gorman C, Harnett JP, Sanders KN, Alvir JM, Cuffel BJ. Findings of a U.S. national cardiometabolic screening program among 10,084 psychiatric outpatients. Psychiatr Serv. 2010 Sep;61(9):892-8. doi: 10.1176/ps.2010.61.9.892. PMID 20810587
- [Background] Colton CW, Manderscheid RW. Congruencies in increased mortality rates, years of potential life lost, and causes of death among public mental health clients in eight states. Prev Chronic Dis. 2006 Apr;3(2):A42. Epub 2006 Mar 15. PMID 16539783
- [Background] Mitchell AJ, Vancampfort D, Sweers K, van Winkel R, Yu W, De Hert M. Prevalence of metabolic syndrome and metabolic abnormalities in schizophrenia and related disorders--a systematic review and meta-analysis. Schizophr Bull. 2013 Mar;39(2):306-18. doi: 10.1093/schbul/sbr148. Epub 2011 Dec 29. PMID 22207632
- [Background] Newcomer JW, Hennekens CH. Severe mental illness and risk of cardiovascular disease. JAMA. 2007 Oct 17;298(15):1794-6. doi: 10.1001/jama.298.15.1794. No abstract available. PMID 17940236
- [Background] Daumit GL, Dickerson FB, Wang NY, Dalcin A, Jerome GJ, Anderson CA, Young DR, Frick KD, Yu A, Gennusa JV 3rd, Oefinger M, Crum RM, Charleston J, Casagrande SS, Guallar E, Goldberg RW, Campbell LM, Appel LJ. A behavioral weight-loss intervention in persons with serious mental illness. N Engl J Med. 2013 Apr 25;368(17):1594-602. doi: 10.1056/NEJMoa1214530. Epub 2013 Mar 21. PMID 23517118
- [Background] Robinson DG, Schooler NR, Correll CU, John M, Kurian BT, Marcy P, Miller AL, Pipes R, Trivedi MH, Kane JM. Psychopharmacological Treatment in the RAISE-ETP Study: Outcomes of a Manual and Computer Decision Support System Based Intervention. Am J Psychiatry. 2018 Feb 1;175(2):169-179. doi: 10.1176/appi.ajp.2017.16080919. Epub 2017 Sep 15. PMID 28945118